CLINICAL TRIAL: NCT07242248
Title: Real World Observation of Guselkumab Treatment in Patients With Ulcerative Colitis and Crohn's Disease - a Study of Treatment Outcomes in the UK
Brief Title: A Study to Observe Real-world Evidence of Guselkumab Treatment in Participants With Ulcerative Colitis and Crohn's Disease in the United Kingdom (UK)
Acronym: GUSTO-UK
Status: Recruiting | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNTO1959IBD4006; CNTO1959IBD4006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease; Colitis, Ulcerative; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Moderate-to-Severe Ulcerative Colitis (UC) or Crohn's Disease (CD): Participants with confirmed diagnosis of moderate-to-severe UC or CD treated with guselkumab as per standard clinical practice will be enrolled. No drug will be provided as part of this study. Only data available from standard clinical practice and medical records will be collected.

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness (how well the treatment works) of Guselkumab, by lines of treatment and subpopulations, and what are the outcomes of treatment (clinical outcomes) in adult participants with moderately to severely active Ulcerative Colitis (UC) or Crohn's Disease (CD) under real-world settings. CD and UC are the main type of Inflammatory bowel disease, a group of inflammatory conditions of the colon and small intestine.

ELIGIBILITY:
Inclusion Criteria:

* Must be eligible for biologic treatment and initiate guselkumab according to the approved indications as described in the current version of the summary of product characteristics (SmPC) of the drug. Decision to prescribe must solely be made by the treating physician in line with the Trust's/ Health Board's treatment guidance. Enrolment must take place before or at the day of first administration (but after treatment decision by physician)
* Must have a confirmed diagnosis of moderate-to-severe Crohn's Disease (CD) or Ulcerative Colitis (UC) recorded in their medical records
* Must sign a informed consent form (ICF) allowing source data verification in accordance with local requirements

Exclusion Criteria:

* Contraindicated to guselkumab per the label
* Is currently enrolled in an interventional clinical study
* Has been previously exposed to interleukin (IL)-23 inhibitors, including Tremfya® (guselkumab), Skyrizi ® (risankizumab) and Omvoh® (mirikizumab). As an exception, participants with history of ustekinumab exposure, may be included
* Has a history of more than 4 lines of advanced inflammatory bowel disease (IBD) therapy (biologics and /or small molecules)
* Is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with confirmed diagnosis of moderate-to-severe Crohn's disease (CD) or Ulcerative colitis (UC) disease.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2029-03-05 (Estimated); Study Completion 2029-03-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Clinical Remission for Crohn's Disease (CD) as Measured by Harvey-Bradshaw Index (HBI) | Up to Week 96
  HBI score is used to assess disease severity and treatment effectiveness. The HBI consists of a 5-part questionnaire, assessing general wellbeing, abdominal pain, number of liquid stools per day, abdominal mass and complications. Clinical remission for CD is defined as the HBI score less than or equal to (<=) 4.
Number of Participants Achieving Clinical Remission for Ulcerative Colitis (UC) as Measured by Partial Mayo Score (PMS) | Up to Week 96
  Mayo scoring system is used to assess disease severity and treatment effectiveness. Clinical remission for UC is defined as the PMS score <=2 and a rectal bleeding subscore of 0.
Number of Participants Achieving Clinical Response for CD as Measured by HBI | Up to Week 96
  HBI score is used to assess disease severity and treatment effectiveness. The HBI consists of a 5-part questionnaire, assessing general wellbeing, abdominal pain, number of liquid stools per day, abdominal mass and complications. Clinical response for CD is defined as the HBI score less than or equal to (<=) 4 or a decrease by greater than or equal to (>=) 3.
Number of Participants Achieving Clinical Response for UC as Measured by PMS | Up to Week 96
  Mayo scoring system is used to assess disease severity and treatment effectiveness. Clinical response for UC is defined as the PMS <4 or >=30 percent (%) reduction of baseline PMS.
Number of Participants Achieving Corticosteroid-free Remission for CD as Measured by HBI | Up to Week 96
  Corticosteroid-free remission for CD is defined as no use of steroids for at least 30 days and HBI score <=4. HBI score is used to assess disease severity and treatment effectiveness.
Number of Participants Achieving Corticosteroid-free Remission for UC as Measured by PMS | Up to Week 96
  Corticosteroid-free clinical remission for UC is defined as no use of steroids for at least 30 days and PMS <2 and a rectal bleeding subscore of 0. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Number of Participants Achieving Corticosteroid-free Clinical Response for CD as Measured by HBI | Up to Week 96
  Corticosteroid-free clinical response for CD is defined as no use of steroids for at least 30 days and a reduction in HBI score by >=3 points from baseline or achieving HBI score <=4. HBI score is used to assess disease severity and treatment effectiveness.
Number of Participants Achieving Corticosteroid-free Clinical Response for UC as Measured by PMS | Up to Week 96
  Corticosteroid-free clinical response for UC is defined as no use of steroids for at least 30 days and PMS <4 or >=30% reduction from baseline. Mayo scoring system is used to assess disease severity and treatment effectiveness.
Number of Participants Achieving Patient-Reported Outcome (PRO)-2 Corticosteroid-Free Remission for CD as Measured by HBI | Up to Week 96
  Participants with corticosteroid-free remission by PRO-2 will be assessed. An abdominal pain (AP) score <=1 and a mean stool frequency (SF) score <=3 and no worsening of AP or SF compared with baseline and no use of corticosteroids for at least 30 days will be defined as a PRO-2 corticosteroid-free remission.
Number of Participants Achieving PRO-2 Corticosteroid-Free Remission for UC as Measured by PMS | Up to Week 96
  Participants with corticosteroid-free remission by PRO-2 will be assessed. An SF score of 0 or 1, where it has not increased from baseline, and a rectal bleeding score of 0 with no use of corticosteroids for at least 30 days will be defined as a corticosteroid-free PRO-2 remission.

SECONDARY OUTCOMES:
Number of Participants with Early Responses to Guselkumab Measured Using PRO-2 Components for UC | Baseline (at Week 0), Weeks 1, 2, 4, 8, 12
  Participants with early responses to guselkumab using PRO-2 components will be assessed and reported via patient diary card.
Number of Participants with Early Responses to Guselkumab Measured Using PRO-2 Components for CD | Baseline (at Week 0), Weeks 1, 2, 4, 8, 12
  Participants with early responses to guselkumab using PRO-2 components will be assessed and reported via patient diary card.
Number of Participants with Early Responses to Guselkumab Measured Using Bowel Urgency | Baseline (at Week 0), Weeks 1, 2, 4, 8, 12
  Participants with early responses to guselkumab using bowel urgency will be assessed and reported via patient diary card. Change in bowel urgency for participants will be asked, that is, how severe were the bowel urgency.
Time to Guselkumab Persistence | Up to Week 96
  Persistence with guselkumab will be measured through time to discontinuation (defined as time at which the next infusion should have taken place for a participant after their last scheduled infusion).
Characteristics of Participants Receiving Guselkumab Treatment: Age | At Baseline
  Characteristics of participants (age) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Sex | At Baseline
  Characteristics of participants (sex) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Previous IBD Medication Use, Smoking Status and History, History of UC and History of CD | At Baseline
  Characteristics of participants (previous IBD medication use, smoking status and history, history of UC and history of CD) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Height | At Baseline
  Characteristics of participants (height) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Weight | At Baseline
  Characteristics of participants (weight) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Disease Severity | At Baseline
  Characteristics of participants (disease severity at index) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Age at Diagnosis | At Baseline
  Characteristics of participants (age at diagnosis) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Disease Duration | At Baseline
  Characteristics of participants (disease duration) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Comorbid Diagnoses | At Baseline
  Characteristics of participants (comorbid diagnoses) receiving guselkumab treatment will be reported.
Characteristics of Participants Receiving Guselkumab Treatment: Previous IBD-Related Surgeries | At Baseline
  Characteristics of participants (IBD-related surgeries) receiving guselkumab treatment will be reported.
Number of Participants with Adverse Events (AEs) | Up to Week 96
  An adverse event is any untoward medical occurrence in a patient administered a medicinal product. An AE does not necessarily have a causal relationship with the treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal finding or lack of expected pharmacological action), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Change in C-reactive protein (CRP) Levels | Baseline up to Week 96
  Change in CRP levels since guselkumab initiation will be reported.
Number of Participants with CRP Normalization | At Week 0, 4, 12, 48 and 96
  Participants with CRP normalization (among participants with CRP elevated at baseline) since guselkumab initiation will be reported.
Change in Faecal Calprotectin (Fcal) Levels | Baseline up to Week 96
  Change in Fcal levels since guselkumab initiation will be reported.
Number of Participants with Fcal Normalization | At Week 0, 4, 12, 48 and 96
  Participants with Fcal normalization (among participants with faecal calprotectin [Fcal] elevated at baseline) since guselkumab initiation will be reported.
Change in Albumin Levels | At Week 0, 4, 12, 48 and 96
  Change in albumin levels to assess anaemia and nutritional status will be reported.
Change in Hemoglobin Levels | At Week 0, 4, 12, 48 and 96
  Change in hemoglobin levels to assess anaemia and nutritional status will be reported.
Change in Platelets Levels | At Week 0, 4, 12, 48 and 96
  Change in platelets levels to assess anaemia and nutritional status will be reported.
Number of Participants Receiving Concomitant IBD Medications During Guselkumab Treatment | Baseline up to Week 96
  Number of participants receiving concomitant medications for UC and CD will be reported.
Health-related Quality of Life (HRQoL) as Measured by Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Scale Score | Baseline (at Week 0), Weeks 12, 48 and 96
  Health related quality of life changes as measured by SIBDQ will be reported. SIBDQ is a 10-item instrument developed to assess the participants perception of their health status specifically related to IBD over the past two weeks. The SIBDQ evaluates the following dimensions: psychological well-being (feelings of emotional health and stability), physical well-being (the impact of disease symptoms on physical health), social function (the influence of the disease on social activities and interactions) and digestive function (the effect of gastrointestinal symptoms on daily life). The total score ranges from 10 (worst health) to 70 (best health).
HRQoL as Measured by Bowel Urgency | Baseline (at Week 0), Weeks 12, 48 and 96
  Health related quality of life changes as measured by bowel urgency will be reported. Change in bowel urgency for participants will be asked, that is, how severe were the bowel urgency.
HRQoL as Measured by PRO-2 Components for Participants with CD | Baseline (at Week 0), Weeks 12, 48 and 96
  PRO-2 components that is change in SF and AP will be reported. Change in SF for participants will be asked, that is, how many bowel movements they had in last 24 hours, how many of those were very soft or liquid, or how many has occurred during the night. Change in AP for participants will be asked, that is, how severe was the abdominal pain in the last 24 hours.
HRQoL as Measured by PRO-2 Components for Participants with UC | Baseline (at Week 0), Weeks 12, 48 and 96
  PRO-2 components that is change in SF and rectal bleeding will be reported. Change in SF for participants will be asked, that is, how many bowel movements they had in last 24 hours, how many of those were very soft or liquid, or how many has occurred during the night. Change in rectal bleeding for participants will be asked, that is, how severe were the rectal bleedings in the last 24 hours.
HRQoL as Measured by IBD-Control Questionnaire (ICHOM) | Baseline (at Week 0), Weeks 12, 24, 48, 72 and 96
  Health related quality of life changes as measured by ICHOM will be reported. ICHOM measures overall disease control from the participants perspective.
Fatigue Measured by Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) Scale | Baseline (Week 0), 12, 48, and 96
  FACIT-F scale is a 13-item instrument that evaluates fatigue/tiredness and its impact on daily activities and functioning in chronic diseases. It includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning (for example, sleeping and social activities) over the last 7 days. The total FACIT-F score ranges from 0 to 52, with a higher score indicating less fatigue.
Number of Participants Achieving Endoscopic Response for Participants with CD as Measured by Simple Endoscopy Score-CD (SES-CD) | Baseline (at Week 0), Weeks 48 and 96
  Endoscopic response is defined as 50% improvement from baseline in SES-CD total score, or SES-CD total score <4.
Number of Participants Achieving Endoscopic Remission for Participants with CD as Measured by SES-CD | Baseline (at Week 0), Weeks 48 and 96
  Endoscopic remission is defined as SES-CD total score <4 with at least 2 points reduction from baseline and no sub-score >1 in any individual component.
Number of Participants Achieving Endoscopic Improvement for Participants with UC as Measured by Mayo Score | Baseline (at Week 0), Weeks 48 and 96
  Endoscopic Improvement is defined as a Mayo score <=1.
Number of Participants Achieving Endoscopic Normalization for Participants with UC as Measured by Mayo Score | Baseline (at Week 0), Weeks 48 and 96
  Endoscopic normalization is defined as a Mayo score =0.
Number of Participants Achieving Histologic Improvement | At Weeks 0, 48 and 96
  Histologic improvement is defined as neutrophil infiltration in <5% of crypts, no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system, that is, Geboes score <=3.1.
Number of Participants Achieving Histologic Remission | At Weeks 0, 48 and 96
  Histologic remission is defined as the absence of neutrophils from the mucosa (both lamina propria and epithelium), no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system, that is, Geboes score <=2B.0.
Number of Participants with CD Achieving Intestinal Ultrasound (IUS) Response | Baseline (at Week 0), Weeks 24, 48, 72, and 96
  IUS Response is defined as reduction of 25% in bowel wall thickness (BWT) or a reduction from baseline of BWT >2 millimeter (mm) or reduction from baseline BWT >1 mm plus a decrease from baseline in color doppler >1 point per baseline pathological segment.
Number of Participants with CD Achieving IUS Remission | Baseline (at Week 0), Weeks 24, 48, 72, and 96
  IUS Remission is defined as BWT <3 mm for ileum and colon plus Color Doppler signal (CDS) 0 in all segments.
Change from Baseline in Satisfaction with Guselkumab Treatment Using Treatment Satisfaction Questionnaire for Medication (TSQM) | Baseline (Week 0), Weeks 12, 48, and 96
  TSQM-9 is an abbreviated version of the 14-item TSQM, and is a reliable and valid measure to assess treatment satisfaction. It consists of 9 items distributed in the domains: side effects, effectiveness, convenience, and global satisfaction, with scores at each domain ranging from 0 to 100. with higher score indicating higher treatment satisfaction.
Change in Number of UC/CD Emergency Room Visits | Baseline, Weeks 12, 48 and 96
  Change in the number of emergency room visits for treatment of UC/CD will be reported.
Change in Number of UC/CD-Hospitalizations | Baseline, Weeks 12, 48 and 96
  Change in the number of hospitalizations for treatment of UC/CD will be reported.
Change in Number of UC/CD Surgeries | Baseline, Weeks 12, 48 and 96
  Change in the number of surgeries for treatment of UC/CD will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Limited Clinical Trial, Study Director — Janssen-Cilag Limited
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No